CLINICAL TRIAL: NCT04322643
Title: A Phase II Study of Intermittent Checkpoint Inhibitor Therapy in Patients With Advanced Urothelial Carcinoma
Brief Title: Intermittent Checkpoint Inhibitor Therapy In Patients With Advanced Urothelial Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI preference
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE6819
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Results first posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — pembrolizumab; atezolizumab; durvalumab; Nivolumab; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CPI therapy (Experimental): Patients will be treated with CPI therapy for at least 24 weeks (+/- 4 weeks) as per standard of care (SOC), at which time those with a tumor burden reduction of 10% or greater will suspend CPI therapy.
  Interventions: Drug: Pembrolizumab; Drug: Atezolizumab; Drug: Durvalumab; Drug: Nivolumab; Drug: Avelumab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg IV over 30 minutes every 3 weeks
  Other Names: KEYTRUDA
Drug: Atezolizumab — Atezolizumab 1200 mg IV over 60 minutes every 3 weeks. (if first dose is tolerated, all subsequent infusions may be delivered over 30 minutes)
  Other Names: TECENTRIQ
Drug: Durvalumab — Durvalumab 10 mg/kg IV over 60 minutes every 2 weeks.
  Other Names: IMFINZI
Drug: Nivolumab — Nivolumab 480mg IV over 30 minutes every 4 weeks
  Other Names: OPDIVO
Drug: Avelumab — Avelumab 800 mg IV over 60 minutes every 2 weeks
  Other Names: BAVENCIO

SUMMARY:
The purpose of this study is to test the safety and effectiveness of immunotherapy (checkpoint inhibitor therapy) in advanced bladder cancer when given intermittently. An unanswered question with the use of CPI (checkpoint inhibitor) is the duration of therapy required for optimal clinical benefit. In the absence of progressive disease or unacceptable toxicities, there are currently no specified criteria for treatment discontinuation. Strategies to reduce toxicity and maximize benefit require investigation. Thus, novel dosing schedules, early discontinuation considerations, and biomarkers of response are needed to identify patients who can sustain disease regression while off of therapy.

DETAILED DESCRIPTION:
A phase II study design to investigate the use of any CPI on an intermittent dosing schedule. Patients with advanced urothelial carcinoma (aUC) who treatment refractory or cisplatin ineligible will receive CPI of choice as per standard dosing. Patients who have initial >/=10% tumor burden reduction will discontinue the CPI until they experience a >/=20% disease progression following 24 weeks +/- 4 weeks of immunotherapy, at which time CPI therapy will be restarted.

All patients who do not meet criteria for the CPI intermittent phase of the study will be treated until unacceptable toxicity or RECIST-defined PD. Patients with RECIST-defined PD may continue CPI therapy at the discretion of the treating MD. These patients will continue with normal imaging every 12 weeks. In cases where a patient is continued on therapy after PD and develops subsequent PD (> 20% increase in sum of target lesions compared to the initial PD tumor measurements, the patient will come off study).

Patients who meet criteria for the intermittent phase (i.e., have >/=10% tumor burden reduction) will not receive CPI therapy. Imaging will continue per protocol (every 12 weeks from the initial date they stopped CPI therapy). Patients who have RECIST defined PD on the intermittent phase should reinitiate CPI therapy. Patients who have a subsequent decrease in tumor burden >/=10% can then restart CPI therapy as per protocol.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age.
* Histological confirmation of urothelial carcinoma (any histology)
* Advanced or metastatic urothelial carcinoma.
* Measurable disease as defined by RECIST 1.1 criteria
* Has received at least 24 weeks (+/- 4 weeks) on CPI therapy per standard of care (SOC) for advanced urothelial carcinoma
* Karnofsky Performance Score (KPS) ≥70% (for more information on KPS, please see: http://www.npcrc.org/files/news/karnofsky_performance_scale.pdf)
* Willing and able to provide informed consent.
* Laboratory criteria for study entry must meet the following criteria:

  * Serum creatinine ≤ 2 x ULN OR CrCl ≥ 30 mL/min (measured or calculated using the Cockcroft-Gault formula).
  * Hb ≥ 8.0g/dL
  * AST and ALT ≤ 3.0 x ULN
  * Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)

Exclusion Criteria:

* History of severe hypersensitivity reaction to any monoclonal antibody.
* Patients are excluded if they have known HIV/AIDS.
* Major surgery (eg, cystectomy) less than 28 days prior to the first dose of study drug.
* Any condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 7 days prior to the first dose of study drug. Inhaled steroids and adrenal replacement steroid doses > 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease.
* Known medical condition (eg, a condition associated with diarrhea or acute diverticulitis) that, in the investigator's opinion, would increase the risk associated with study participation or study drug administration or interfere with the interpretation of safety results.
* Pregnant women are excluded from this study because animal studies have demonstrated that PD-1/PD-L1 inhibitors can cause fetal harm when administered to pregnant women. Breastfeeding women are excluded from this study because PD-1/PD-L1 inhibitors may be excreted in human milk and the potential for serious adverse reactions in nursing infants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-03-23 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2023-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Ornstein, MD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Summary results are shared in publications

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CPI Therapy
Started | 4
Completed | 0
Not Completed | 4
Not completed — Study halted prematurely therefore treatment halted. | 4

BASELINE CHARACTERISTICS:
Arm/Group | CPI Therapy
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Sustain a Response Post CPI Suspension
Description: Efficiency, as measured by number of participants that sustain a response post CPI suspension. Response is defined as tumor burden reduction of 10% or greater. Response is measured based on RECIST criteria version 1.1. RECIST 1.1 responses include Complete Response (CR) which is defined as disappearance of all lesions and pathologic lymph nodes; Partial Response (PR) defined as ≥ 30% decrease SLD, no new lesions, no progression of non-target lesions; Stable disease (SD) which is defined as no partial or complete responses; or Progressive disease (PD) defined as ≥ 20% increase SLD compared to smallest SLD in study, or progression of non-target lesions, or new lesions.
Time Frame: At 36 weeks post CPI suspension
Population: All four participants sustained a response after CPI therapy, but this study was terminated prematurely due to the changes in treatment landscape of advanced urothelial carcinoma.
Measure: Count of Participants; unit: Participants
Arm/Group | CPI Therapy
Number analyzed (Participants) | 4
Participants | 4

2. Secondary Outcome: Median Treatment Free Interval (TFI) in Weeks
Description: Median and range TFI in months. Participants will be treated with CPI therapy for at least 24 weeks (+/- 4 weeks) as per standard of care (SOC), at which time those with a tumor burden reduction of 10% or greater will suspend CPI therapy. Participants with a documented increase in ≥ 20% tumor burden (RECIST 1.1 PD) will re-initiate CPI. For those patients who continue to have response, they will remain off therapy.
Time Frame: Up to 36 weeks from end of treatment, through study completion an average of 160 weeks
Population: Due to slow accrual and premature trial closure, data were incompletely collected and not analyzed, with no plans for future analysis. The true participant TFI is not available as this study terminated prematurely and ended follow up period. The outcome measure data is based on TFI at time of termination.
Measure: Median (Full Range); unit: weeks
Arm/Group | CPI Therapy
Number analyzed (Participants) | 4
weeks | 94.1 [36.1 to 106.8]

3. Secondary Outcome: Overall Response Rate (ORR)
Description: Response to re-initiation of CPI therapy as measured by overall response rate (ORR) defined as the percentage of participants who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) as assessed by RECIST 1.1
Time Frame: Up to 36 weeks from end of treatment, through study completion an average of 160 weeks
Population: Due to slow accrual and premature trial closure, data were incompletely collected and not analyzed, with no plans for future analysis. All four participants sustained a response after CPI therapy, but this study was terminated prematurely due to the changes in treatment landscape of advanced urothelial carcinoma.
Measure: Count of Participants; unit: Participants
Arm/Group | CPI Therapy
Number analyzed (Participants) | 4
Participants
  Partial Response | 4
  Complete Response | 0
  Stable Disease | 0
  Progressive Disease | 0

4. Secondary Outcome: Number of Participants With Progression Free Survival (PFS)
Description: Progression free survival (PFS) defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first as assessed by RECIST 1.1 criteria. PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm and the appearance of ≥1 new lesions is also considered PD.
Time Frame: Up to 36 weeks from end of treatment, through study completion an average of 160 weeks
Population: 4/4 patients remained progression-free survival at the time of study termination.
Measure: Count of Participants; unit: Participants
Arm/Group | CPI Therapy
Number analyzed (Participants) | 4
Participants | 4

5. Secondary Outcome: Number of Participants With Overall Survival (OS)
Description: Overall Survival (OS) defined as the time from randomization to death due to any cause
Time Frame: Up to 36 weeks from end of treatment, through study completion an average of 160 weeks
Population: 4/4 participants were alive at the time of study termination.
Measure: Count of Participants; unit: Participants
Arm/Group | CPI Therapy
Number analyzed (Participants) | 4
Participants | 4

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from beginning study until study completion, and for a minimum of 30 days following the last dose of study treatment; up to 160 weeks, treatment lasted an average of 24 weeks.
Arm/Group | CPI Therapy
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
This study was terminated prematurely due to low enrollment and the changes in the treatment landscape of advanced urothelial carcinoma. Due to premature trial closure, data were incompletely collected and analyzed. There are no plans for future analysis. The outcome measure data is only based on the information that was collected for four participants at the time of study termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT04322643/Prot_SAP_000.pdf
  • Informed Consent Form (2020-02-26): https://cdn.clinicaltrials.gov/large-docs/43/NCT04322643/ICF_001.pdf